CLINICAL TRIAL: NCT02816853
Title: A Randomized, Placebo- and Positive-Controlled, Multiple-Dose, 4-Way Crossover Study to Evaluate the Effects of Domperidone on Cardiac Repolarization in Chinese Healthy Subjects
Brief Title: Study to Evaluate the Effects of Domperidone on Cardiac Repolarization in Chinese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108170; R033812DYP1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-06-03; First posted 2016-06-29 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Domperidone; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): Participants will be randomly assigned to 1 of 4 treatment sequence groups based on a computer generated randomization schedule and will receive the following 4 treatments in order specified by randomization: Treatment A (1 domperidone 10 mg tablet 3 times a day (tid) + 1 placebo tablet tid on Days 1 to 3 and a single dose of 1 domperidone 10 mg tablet +1 placebo tablet in the morning of Day 4), Treatment B (2 domperidone 10 mg tablets tid on Days 1 to 3 and a single dose of 2 domperidone 10 mg tablets in the morning of Day 4), Treatment C (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets in the morning of Day 4) and Treatment D (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets + 1 moxifloxacin 400 mg tablet in the morning of Day 4).
  Interventions: Drug: Domperidone; Drug: Placebo; Drug: Moxifloxacin
- Sequence 2 (Experimental): Participants will be randomly assigned to 1 of 4 treatment sequence groups based on a computer generated randomization schedule and will receive the following 4 treatments in order specified by randomization: Treatment A (1 domperidone 10 mg tablet 3 times a day (tid) + 1 placebo tablet tid on Days 1 to 3 and a single dose of 1 domperidone 10 mg tablet +1 placebo tablet in the morning of Day 4), Treatment B (2 domperidone 10 mg tablets tid on Days 1 to 3 and a single dose of 2 domperidone 10 mg tablets in the morning of Day 4), Treatment C (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets in the morning of Day 4) and Treatment D (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets + 1 moxifloxacin 400 mg tablet in the morning of Day 4).
  Interventions: Drug: Domperidone; Drug: Placebo; Drug: Moxifloxacin
- Sequence 3 (Experimental): Participants will be randomly assigned to 1 of 4 treatment sequence groups based on a computer generated randomization schedule and will receive the following 4 treatments in order specified by randomization: Treatment A (1 domperidone 10 mg tablet 3 times a day (tid) + 1 placebo tablet tid on Days 1 to 3 and a single dose of 1 domperidone 10 mg tablet +1 placebo tablet in the morning of Day 4), Treatment B (2 domperidone 10 mg tablets tid on Days 1 to 3 and a single dose of 2 domperidone 10 mg tablets in the morning of Day 4), Treatment C (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets in the morning of Day 4) and Treatment D (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets + 1 moxifloxacin 400 mg tablet in the morning of Day 4).
  Interventions: Drug: Domperidone; Drug: Placebo; Drug: Moxifloxacin
- Sequence 4 (Experimental): Participants will be randomly assigned to 1 of 4 treatment sequence groups based on a computer generated randomization schedule and will receive the following 4 treatments in order specified by randomization: Treatment A (1 domperidone 10 mg tablet 3 times a day (tid) + 1 placebo tablet tid on Days 1 to 3 and a single dose of 1 domperidone 10 mg tablet +1 placebo tablet in the morning of Day 4), Treatment B (2 domperidone 10 mg tablets tid on Days 1 to 3 and a single dose of 2 domperidone 10 mg tablets in the morning of Day 4), Treatment C (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets in the morning of Day 4) and Treatment D (2 placebo tablets tid on Days 1 to 3 and a single dose of 2 placebo tablets + 1 moxifloxacin 400 mg tablet in the morning of Day 4).
  Interventions: Drug: Domperidone; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Domperidone — Domperidone 10 mg or 20 mg tablets will be administered.
Drug: Placebo — Matching placebo will be administered.
Drug: Moxifloxacin — Moxifloxacin 400 mg tablet will be administered.

SUMMARY:
The purpose of this study is to assess the effects of domperidone on the QTc interval duration in Chinese healthy adult participants after multiple domperidone doses of 10 milligram (mg) 3 times a day (tid) and 20 mg tid.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. This determination must be recorded in the participants source documents and signed by the investigator
* Participant must be healthy on the basis of clinical laboratory tests performed at Screening. If the results of the serum chemistry panel including liver enzymes, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participants source documents and signed by the investigator
* A woman, must have been proved to be non-pregnant via a highly sensitive serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at Screening; and a negative urine pregnancy test on Day -1 of each treatment period
* Due to the lack of adequate reproductive toxicity data, in addition to the user independent highly effective method of contraception, a male or female condom with or without spermicide is required. Male condom and female condom should not be used together (due to risk of failure with friction)
* Body mass index (BMI; weight [kilogram {kg}]/height^2 [meter {m}]^2) between 18 and 30 kilogram per meter square [kg/m^2] (inclusive), and body weight not less than 50 kilogram (kg)

Exclusion Criteria:

* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, gastro-intestinal disease, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Presence of hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia
* Clinically significant abnormal physical examination, vital signs or 12-Lead electrocardiogram (ECG) at Screening or at admission to the study center as deemed appropriate by the investigator
* Known allergy to the Domperidone or any of the excipients of the formulation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in QTc Interval Based on Fridericia Correction Method (QTcF) | Baseline, Day 1 and Day 4
  The QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by electrocardiograms (ECG).

SECONDARY OUTCOMES:
Change From Baseline in QTc Interval Based on Study-Specific Power Correction (QTcP) | Baseline, Day 1 and Day 4
  The QT interval corrected for heart rate (QTc interval) using study-specific power correction method will be measured by electrocardiograms (ECG).
Change From Baseline in QTc Interval Based on Bazett Method (QTcB) | Baseline, Day 1 and Day 4
  The QT interval corrected for heart rate (QTc interval) using Bazett method will be measured by electrocardiograms (ECG).
Change From Baseline in HR, QRS and PR Intervals | Baseline, Day 4
  The HR, QRS, and PR Intervals will be measured by ECG.
Maximum Observed Plasma Concentration | Day 1
  The Cmax is the maximum observed plasma concentration.
Time to Reach the Maximum Plasma Concentration (Tmax) | Day 1 and Day 4 (Predose up to 5 hours post dose)
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve During the First Dosing Interval (AUCtau) | Day 1 and Day 4 (Predose up to 5 hours post dose)
  The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Maximum Plasma Concentration at Steady State (Cmax,ss) | Day 4 (Predose up to 5 hours post dose)
  The Cmax,ss is the maximum observed plasma concentration at steady state.
Minimum Plasma Concentration at Steady State (Cmin,ss) | Day 4 (Predose up to 5 hours post dose)
  The Cmin,ss is the minimum observed plasma concentration at steady state.
Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) as a Measure of Safety and Tolerability | Up to End of Study (4 to 10 days after last study drug administration)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Beijing, China